CLINICAL TRIAL: NCT04764682
Title: Determining Molecular Drivers of Radiation Dermatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Laura A. Vallow, Principal Investigator, Mayo Clinic
Other Study IDs: 19-005445
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin tissue. A 3mm punch biopsy will be collected at the time of surgery and during the final week of radiation treatment. One half of the sample will be placed in a separate cryovial container RNA later and the other half will be placed in a cryovial and flash frozen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is being conducted to address key gaps in current knowledge and set the stage for rational design of strategies to prevent (pre-exposure to radiation), mitigate (post-exposure to radiation before overt signs/symptoms appear), and/or treat (post-onset of signs/symptoms) radiation dermatitis (itchy, dry skin or a rash on swollen, reddened skin).

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving standard-of-care postoperative radiation therapy (2-2.7 Gy per fraction) to the breast and/or chest wall for breast cancer treatment.
* Tissue diagnosis of breast cancer.
* Age > 18 years
* Signed informed consent.
* Complete blood count within normal limits within the preceding 2 weeks.

Exclusion criteria:

* Induction chemotherapy or biologic therapy
* Concurrent chemotherapy or biologic therapy
* Autoimmune disease with skin manifestations - psoriasis, dermatomyositis, scleroderma, eczema, polymyositis
* Allergy to lidocaine anesthesia
* Known bleeding diathesis (anticoagulation with warfarin, coagulation/bleeding disorders, vitamin C or K deficiency, thrombocytopenia)
* History of keloids or easy scarring

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women aged 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in skin | Baseline, final week of radiation
  A skin punch biopsy will be obtained from a visible area of skin that harbors signs of clinical radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vallow, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20509173